CLINICAL TRIAL: NCT06668870
Title: Electronic Health Record-Integrated Patient-Generated Data to Support Clinical Care and Research
Brief Title: Electronic Health Record-Integrated Patient-Generated Data
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00113850; 1UM1TR004929-01 (NIH)
Record Dates: First submitted 2024-10-28; First posted 2024-11-01 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-09

CONDITIONS: Sepsis
Keywords: patient-generated data collection; electronic health record monitoring; transitional care
MeSH Terms: conditions — Sepsis | interventions — Educational Status; Patient Generated Health Data

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supportive Messaging (Experimental): Supportive messaging is a behavioral intervention delivered to motivate patients to engage with targeted patient-generated data collection tools. Participants will be asked to complete patient-generated data. At baseline, all patients will receive education about the collection of patient-generated data, training in using the data collection tools, and guidance on the standard frequency for collection and sharing of information. At baseline and regular intervals throughout follow up, the supportive messaging arm will receive added text messaging to engage patients and deliver personalized reminders to complete monitoring tasks.
  Interventions: Behavioral: Supplemental Text Messaging
- No Supportive Messaging (Active Comparator): Participants will be asked to complete patient-generated data. At baseline, participants will receive education about the collection of patient-generated data, training in using the data collection tools, and guidance on the standard frequency for collection and sharing of information. Participants will not receive added text messaging to engage patients and deliver personalized reminders to complete monitoring tasks.
  Interventions: Behavioral: Education and Training for Patient-Generated Data

INTERVENTIONS:
Behavioral: Supplemental Text Messaging — Will receive education about the collection of patient-generated data, training in using the data collection tools, and guidance on the standard frequency for collection and sharing of information. Supplemental text messages will be sent to engage patients and deliver personalized reminders to complete monitoring tasks.
  Arms: Supportive Messaging
Behavioral: Education and Training for Patient-Generated Data — Will receive education about the collection of patient-generated data, training in using the data collection tools, and guidance on the standard frequency for collection and sharing of information.
  Arms: No Supportive Messaging

SUMMARY:
The purpose of this study is to find out if patients that receive supportive messaging with response adaptation are more likely to adhere to patient-generated data collection and electronic health record integration, compared to patients that do not receive supportive messaging.

DETAILED DESCRIPTION:
This project will directly inform re-usable strategies to support the integration of important patient-generated data (PGD) into the electronic health record to improve clinical care and research. For this application, investigators propose to develop and test the PGD translational science innovation in patients recovering from sepsis. This diverse patient population frequently suffers from long-term complications that are ideally suited for development and demonstration of strategies to collect, integrate, and examine PGD and builds directly on the study team's robust research portfolio on improving sepsis recovery.

ELIGIBILITY:
Inclusion Criteria:

* Discharged alive from the hospital without hospice care who meet clinical criteria for infection and organ dysfunction consistent with sepsis
* Enrolled into the Sepsis Transition and Recovery program
* Enrolled or willing to enroll as an Epic MyChart user

Exclusion Criteria:

* Discharged from the hospital with hospice care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Proportion of Completed Versus Requested Patient-Generated Data | 90 days post hospital discharge
  Patient generated data completion defined as the proportion of completed vs requested patient generated data elements.

SECONDARY OUTCOMES:
Number of Readmissions | 90 days post hospital discharge
  Number of readmissions to inpatient or observation status due to any cause assessed via electronic health record.
Number of Deaths | 90 days post hospital discharge
  Number of participant deaths due to any cause, assessed via electronic health record and national data sources integrated in the enterprise data warehouse.
Number of Emergency Department Visits | 90 days post hospital discharge
  Number of Emergency Department visits assessed via electronic health record.
Number of Outpatient Clinic Visits | 90 days post hospital discharge
  Number of outpatient clinic visits assessed via electronic health record
Number of Hospital-Free Days | 90 days post hospital discharge
  Number of hospital-free days calculated by total of days alive minus days hospitalized, measured from electronic health record data.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Kowalkowski, PhD, Principal Investigator — Atrium Health Wake Forest Baptist

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification will be shared (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Will share with researchers who provide a methodologically sound proposal to assist in achieving aims in the approved proposal. Proposals should be directed to ehale@wakehealth.edu. To gain access, data requestors will need to sign a data access agreement.